CLINICAL TRIAL: NCT07076940
Title: The Effect of Mindfulness-Based Education on Stress Perception and Well-Being in Caregivers of Individuals Diagnosis With Schizophrenia
Brief Title: Mindfulness-Based Education for Caregivers of Individuals Diagnosis With Schizophrenia
Acronym: MBECIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Azize Gözde Atakoğlu, Principal Investigator, PhD Student, Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25.05.2022 / 90
Record Dates: First submitted 2025-07-10; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Mindfulness; Mindfulness Based Stress Reduction; Caregivers; Stress Perception; Psychological Well-being; Schizophrenia Disorder
Keywords: Mindfulness; Caregivers; Stress perception; Psychological well-being; Schizophrenia
MeSH Terms: conditions — Psychological Well-Being; Schizophrenia

STUDY DESIGN:
Intervention Model Description: The study included the "Mindfulness Group (n: 15), "Psychoeducation Group (n: 15)," and control group (n: 30). Different patient relatives were randomly assigned to each group. The mindfulness group received five sessions (one day per week, 60 minutes, for a total of five consecutive weeks). The psychoeducation group completed a "Psychoeducation Program" themed around stress, well-being, and mindfulness in two sessions (two sessions over five weeks, each session lasting 60 minutes). The control group received no intervention. Posttest measurements (n: 30) were taken after the completion of the training program for the mindfulness and psychoeducation groups. Follow-up tests (n: 30) were conducted simultaneously with the mindfulness and psychoeducation groups one month later.
Who Masked: Participant
Masking Description: Participants were assigned to different groups. Intervention plans were made for each group on different days to minimize contact between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness Group (Experimental): The mindfulness-based training program was completed in a total of five sessions (one day per week, 60 minutes, for a total of five consecutive weeks).
  Interventions: Other: Mindfulness-based Training Program
- Psychoeducation Group (Other): The "Psychoeducational Program," themed around stress, well-being, and mindfulness, was completed in two sessions (two sessions over five weeks, each lasting 60 minutes).
  Interventions: Other: Psychoeducational Program
- Control Group (No Intervention): No intervention was administered.

INTERVENTIONS:
Other: Mindfulness-based Training Program — The mindfulness-based training program was completed in a total of five sessions (one day per week, 60 minutes, for a total of five consecutive weeks).
  Arms: Mindfulness Group
Other: Psychoeducational Program — The "Psychoeducational Program," themed around stress, well-being, and mindfulness, was completed in two sessions (two sessions over five weeks, each lasting 60 minutes).
  Arms: Psychoeducation Group

SUMMARY:
The research is carried out by PhD student Azize Gözde Atakoğlu under the supervision of Associate Professor Gülcan Kendirkıran.

This study was conducted with a randomized control group, experimental research design in order to determine the effects of mindfulness-based training on stress perception and well-being in caregivers of individuals diagnosed with schizophrenia. The research data were collected at the Community Mental Health Center affiliated with a Training and Research Hospital in Istanbul between 15 September 2022 and 1 February 2023. Before commencing the study, an ethical approval decision was obtained from the Haliç University Non-Interventional Clinical Research Ethics Committee (May 25, 2022-90). Subsequently, an institutional permit for the study (June 28, 2022-637) was obtained from the Istanbul Provincial Health Directorate Bakırköy Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital, along with the ethics committee approval. The sample of the study consisted of caregivers of individuals diagnosed with schizophrenia, 15 in the intervention group, 15 in the psychoeducation group, and 30 in the control group (n=60). The study data were collected using the Personal Information Form, Perceived Stress Scale (PSS), Psychological Well-Being Scale (PWS), Participant Experience Form (PEF), Post-Experience Stress Assessment Questionnaire (PSSQ), and Home Application Note Form. Frequency tables and descriptive statistics were used in the interpretation of the findings. For measurement values suitable for normal distribution, "ANOVA" test (F-table value), "Repeated Measures" test (F-table value), for measurement values not suitable for normal distribution, Kruskal-Wallis H" test (χ2-table value), "Friedman" test (χ2-table value) method was used. "Pearson-χ2" was used to examine the relationships between two qualitative variables, and "Spearman" correlation coefficient was used to examine the relationships between two quantitative variables not having normal distribution. As a result of this study, it was found that mindfulness-based intervention reduced stress in caregivers and contributed to psychological well-being (p<0.05). In addition, it was observed that the effect continued even though it decreased in follow-up tests. In this direction, it is recommended that follow-up tests be kept longer and intermediate interventions be added in other studies to be conducted. It is also recommended that qualitative studies be conducted on this subject in order to obtain detailed feedback on the processes related to the initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* The patient they are caring for must have been diagnosed with schizophrenia according to the DSM-V (Diagnostic and Statistical Manual of Mental Disorders) classification at least one year ago
* Living together in the same house for at least one year
* Being directly responsible for the patient's treatment arrangements and care
* Being open to communication and collaboration.

Exclusion Criteria:

* Having any condition that may prevent them from receiving education.
* Having a vision, hearing, or comprehension problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | Before the intervention, immediately after the intervention, and 1 month after the last measurement
  The scale consists of 14 items in a 5-point Likert type. 7 items with positive expressions (4, 5, 6, 7, 9, 10, 13) are reverse coded and high scores indicate a high level of perceived stress. The scale has 2 sub-dimensions as "perception of inadequacy" and "perception of stress/discomfort." The score to be obtained from PSS-14 varies between 0 and 56. The Cronbach's Alpha coefficient of the Turkish scale was determined as 0.84 and its reliability as 0.87. Cronbach's Alpha values obtained in this study are as follows in the whole sample; inadequate self-efficacy perception is 0.89, stress discomfort perception is 0.79, PSS total is 0.89.
Psychological Well-Being Scale | Before the intervention, immediately after the intervention, and 1 month after the last measurement
  The items of PWB are answered on a scale of 1-7, from strongly disagree (1) to strongly agree (7). All items are expressed positively. Scores range from 8 (if strongly disagree is answered to all items) to 56 (if strongly agree is answered to all items). A high score indicates that the person has many psychological resources and strengths. Although the scale does not provide separate measurements of aspects of well-being, it provides an overview of positive functions in different areas that are believed to be important. The Cronbach's alpha internal consistency coefficient obtained in the reliability study of the scale was calculated as .80 (Telef, 2013). Cronbach's Alpha values obtained in this study; is 0.91 in the entire sample.

SECONDARY OUTCOMES:
Personal Information Form | Before the intervention
  This form consisted of 23 multiple-choice and open-ended questions regarding the participants' individual characteristics, their knowledge of caregiving, and their perceptions of mental health-related stress and well-being. The form was developed by the researchers based on literature. Expert opinion was obtained to determine its appropriateness.
Participant Experience Form | Immediately after the intervention
  This form was developed by researchers to identify the experiences of mindfulness group members participating in a mindfulness-based training program, including their emotions, thoughts, and perceptions, as well as their subjective evaluations of the training process. The form consists of nine items, with responses ranging from 1 to 5, from not at all (1) to completely (5).

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan KENDİRKIRAN, Associate Professor, Study Director — Halic University
Locations (1):
- Zeytinburnu Community Mental Health Center, affiliated with the Istanbul Bakırköy Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital., Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No